CLINICAL TRIAL: NCT04807127
Title: A Single-cell Approach to Identify Biomarkers of Pulmonary Toxicity for Immune Checkpoint Blockade
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S63357
Record Dates: First submitted 2021-03-10; First posted 2021-03-19 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Pneumonitis, Interstitial; Immunotherapy; Immune-related Adverse Events
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — Immune Checkpoint Inhibitors; pembrolizumab; durvalumab; Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * BAL samples will not be retained
  * PBMC samples will be stored at -80°C, for batch processing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ICI-pneumonitis: Cancer patients experiencing ICI-pneumonitis
  Interventions: Drug: Immune checkpoint blockade
- Radiotherapy induced pneumonitis: Cancer patients experiencing RT-pneumonitis
  Interventions: Radiation: Radiotherapy
- TKI-induced pneumonitis: Cancer patients experiencing TKI-induced pneumonitis
  Interventions: Drug: Targeted therapy

INTERVENTIONS:
Drug: Immune checkpoint blockade — ICI, administered as standard-of-care treatment
  Other Names: Pembrolizumab; Durvalumab
  Groups: ICI-pneumonitis
Drug: Targeted therapy — TKI, administered as standard-of-care treatment
  Other Names: TKI
  Groups: TKI-induced pneumonitis
Radiation: Radiotherapy — RT, administered as standard-of-care treatment
  Groups: Radiotherapy induced pneumonitis

SUMMARY:
The main goal of this prospective non-interventional exploratory monocentric study is to characterize the immune cell composition of bronchoalveolar lavage (BAL) fluid from cancer patients experiencing cancer therapy-induced pneumonitis on a single-cell scale. These mechanistic insights can directly lead to putative diagnostic biomarkers and therapeutic targets.

A second highly clinically relevant hypothesis is that single-cell profiling of blood samples will reveal circulating biomarkers of ICB toxicity, making non-invasive diagnosis feasible.

DETAILED DESCRIPTION:
The investigators will apply single cell RNA- and TCR-sequencing on up to 5,000 single cells per sample. Additionally, cell surface protein expression can be integrated with the transcriptional information. Various bioinformatics pipelines, including Seurat, will be used to identify different cell clusters, which through marker gene expression will be assigned to known cell types, cellular subtypes or phenotypes. For instance, this will make it possible to monitor the abundance of PD-1/PD-L1 expressing T-cells, cytotoxic T-cells, immune-suppressive myeloid cells etc. The following parameters at single-cell level will be relevant, amongst others:

* The composition and relative abundancies of established immune cell types (e.g. T cells (CD4+, CD8+ and regulatory subsets), NK cells, B cells, MDSCs, macrophages, neutrophils, dendritic cells). Transcriptomic data for each of these immune cell subtypes will be analyzed, allowing characterization of specific gene expression programs that define specific phenotypic states.
* Composition of all stromal cellular subtypes identified by single-cell transcriptomics.
* A gene regulatory network for each cell type and cellular subtype (or cell state) will be established and master transcriptional regulators will be identified. Individual T-cells and T-cell subclusters will be classified based on interferon activation, high rates of proliferation and transcription and increased granzyme expression, which are all indicative of T-cell activation.

Blood samples will be subjected to similar single-cell experimental procedures. First, peripheral blood mononuclear cells (PBMC) are isolated using Ficoll density gradient centrifugation. Single-cell transcriptome analysis in combination with CITE-seq will be performed on 5000 PBMC. Cellular composition will be determined using the same bioinformatic pipelines as used for processing the BAL fluid cells.

ELIGIBILITY:
Inclusion criteria:

* Adult M/F/X (>= 18 years)
* Patients receiving or having received treatment per guidelines
* Patients undergoing bronchoscopy with BAL, for possible cancer treatment-induced pneumonitis
* Not included in other clinical trials
* Signed informed consent form

Exclusion criteria:

• Collected material not suitable for further processing in this study (e.g. bad quality). This decision will be made in consultation with a lab technician and/or bio-informatician, specialized in single-cell analysis.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients experiencing cancer-treatment induced pneumonitis, undergoing bronchoscopy with BAL
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Immune cell proportions, as determined by scRNA-seq, present in ICI-/RT-/TKI-induced pneumonitis BAL fluid | From date of inclusion until study completion, on average 2 years
  By identifying and statistically comparing the percentages of immune cell subtypes present in ICI-/RT-/TKI-induced pneumonitis BAL fluid, we aim to i) understand which immune processes drive these adverse events ii) identify putative molecular biomarkers iii) identify putative therapeutic targets
Differentially expressed genes in BAL fluid, as determined by scRNA-seq, discriminating ICI-/RT-/TKI-induced pneumonitis | From date of inclusion until study completion, on average 2 years
  By identifying differentially expressed genes in ICI- vs. RT- vs. TKI-induced pneumonitis BAL fluid, we aim to i) understand which immune processes drive these adverse events ii) identify putative molecular biomarkers iii) identify putative therapeutic targets

SECONDARY OUTCOMES:
Immune cell proportions, as determined by scRNA-seq, present in ICI-/RT-/TKI-induced pneumonitis peripheral blood mononuclear cells | From date of inclusion until study completion, on average 2 years
  By identifying and statistically comparing the percentages of immune cell subtypes present in ICI-/RT-/TKI-induced pneumonitis peripheral blood mononuclear cells, we aim to i) understand which immune processes drive these adverse events ii) identify putative molecular biomarkers iii) identify putative therapeutic targets
Differentially expressed genes in PBMC, as determined by scRNA-seq, discriminating ICI-/RT-/TKI-induced pneumonitis | From date of inclusion until study completion, on average 2 years
  By identifying differentially expressed genes in ICI- vs. RT- vs. TKI-induced pneumonitis PBMC, we aim to i) understand which immune processes drive these adverse events ii) identify putative molecular biomarkers iii) identify putative therapeutic targets

CONTACTS AND LOCATIONS:
Overall Officials: Els Wauters, MD, PhD, Principal Investigator — University Hospitals - KU Leuven
Locations (1):
- Universitaire Ziekenhuizen Leuven, Leuven, Flemish Brabant, Belgium